CLINICAL TRIAL: NCT04986800
Title: PROACTIVE Parent: Providing Access To Innovative & Evidence-Based Intervention
Brief Title: Providing Access To Innovative & Evidence-Based Intervention
Acronym: PROACTIVE
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Was never funded. Through rounds of grant applications, the intervention changed substantially based on reviewer feedback and feasibility
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Heather Risser, Assistant Professor, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU00214486
Record Dates: First submitted 2021-05-24; First posted 2021-08-03 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Mental Health Issue

STUDY DESIGN:
Intervention Model Description: A service delivery model and telehealth methodology to deliver a combination of mental health evaluation of the child, motivational interviewing, transdiagnostic and evidence-based skills training (ST), and parent training (PT) to parents.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Group (Experimental): Participants in the Intervention Group will receive up to 10 sessions of the PROACTIVE Parent intervention.
  Interventions: Behavioral: PROACTIVE Parent

INTERVENTIONS:
Behavioral: PROACTIVE Parent — PROACTIVE Parent will educate parents about their child's mental health symptoms and treatment, how to talk to the child's therapist to support treatment goals at home and in the community. PROACTIVE Parent will teach parents the function of child behavior, the role of symptomatology in child behaviors, and strategies to promote effective behavior management and healthy coping. Parents will also learn skills to manage their own emotional dysregulation to promote calm parental responding and promote healthy parent-child interaction and communication.

SUMMARY:
PROACTIVE Parent is an educational program designed to improve parenting skills to more effectively manage child behavior and social and emotional needs in children with depressive symptoms. PROACTIVE Parent (Providing Access To Innovative & Evidence-Based Intervention) is a new service delivery model that uses telehealth methodology to engage parents in managing their child's mental health needs. PROACTIVE Parent aims to provide parents with information about their child's mental health symptoms and diagnosis, options for evidence-based treatment interventions, and a free, online application for identifying appropriate and accessible treatment options. PROACTIVE Parent is also designed to provide parents a deeper understanding of the function of child behavior, and strategies to promote effective behavior management and healthy coping. Parents will also learn skills to manage their own emotional dysregulation to promote calm parental responding and healthy parent-child interaction and communication. The investigators will assess the acceptability, feasibility, and preliminary effectiveness of a 10-week curriculum. Outcomes include parent reports of acceptability, utility, feasibility of program elements, and the preliminary effectiveness of the program in improving parent activation, parent empowerment, parent emotion dysregulation, and reducing child mental health and behavioral symptoms, and barriers to treatment participation.

DETAILED DESCRIPTION:
PROACTIVE Parent is an educational program designed to improve parent knowledge, capacity and confidence to more effectively manage child behavior and social and emotional needs in children with depressive symptoms. PROACTIVE Parent (Providing Access To Innovative & Evidence-Based Intervention) is a new service delivery model that uses telehealth methodology to educate parents about their child's mental health (MH) symptoms and treatment, teach parents skills to promote a safe, regulated environment for their youth, and teach parents how to work with their child's therapists to support treatment goals at home and in the community. PROACTIVE Parent will teach parents the function of child behavior, the role of symptomatology in child behaviors, and strategies to promote effective behavior management and healthy coping. Parents will also learn skills to manage their own emotional dysregulation to promote calm parental responding and promote healthy parent-child interaction and communication.

The PROACTIVE Parent model is ideally suited to promote parent's active management of child MH care. Children depend on parents to navigate a complex system of care and support children's coping in the home and community. However, parents may not know how to navigate appropriate treatments, how to communicate with their child's therapist to support treatment goals in the home, or how to interact with their child in a way that supports positive mental health outcomes. These parents require a service model that builds parent capacity to manage their child's MH care. The conceptual framework for the proposed work draws on the concept of parent activation and engagement in their child's MH care, and regulating affect. Activation refers to the parent's knowledge, capacity, and commitment to manage their child's MH care. Engagement refers to actions parents take to manage their child's care. Emotion regulation skills help parents to manage their affect, to engage in calm responding to children's needs and assist children in regulating affect.

PROACTIVE Parent is delivered in weekly 30-minute telehealth coaching sessions over the course of 10 weeks. Parent coaches use motivational interviewing and psychoeducation to improve parent activation and management of their child's MH care. Parent coaches provide parent-training and evidence-based skills training to promote effective parent behavior, healthy coping, and positive parent-child interaction. The parent coach will deliver the PROACTIVE Parent model via telehealth with supplemental online resources, using a publically available service referral system to connect parents to evidence-based treatments and MH providers if needed.

The investigators will recruit Foster Parents of youth in care aged 8 - 13 years, with symptoms or history of depression to examine acceptability, feasibility and preliminary effectiveness of the PROACTIVE Parent program.

The Aims of this project include an open trial, and exploration of the relationship between parent activation and youth MH outcomes.

Aim 1: Conduct a pilot study to test acceptability, utility, feasibility, and preliminary effectiveness. The primary outcomes include: 1) Acceptability, 2) Usefulness, and 3) Feasibility (all measured by post-session questions and post-intervention Customer Satisfaction Survey; Feasibility will also include number of people referred who meet eligibility, number of parents who enroll after referral, time to complete assessments). Aim 2: Assess the preliminary effectiveness of the model to improve parent activation, and empowerment. Aim 3: Assess the preliminary effectiveness to reduce the number, severity, and frequency of child MH symptoms and maladaptive behaviors. Aim 4: Assess preliminary effectiveness of improving parent scores on the DERS and barriers to treatment participation.

If the PROACTIVE Parent model demonstrates feasibility and effectiveness, it could serve as a model for scaling up to a population-based approach to MH treatment for all children.

ELIGIBILITY:
Inclusion Criteria

* Foster parent of child aged 8 - 13 years old with mental health symptoms
* Has access to a device and internet to allow videoconferencing or phone coaching

Exclusion Criteria

* Not currently parenting a child with symptoms or history of depression
* Does not speak English
* Does not have access to a device and internet to allow videoconferencing or phone coaching

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2024-12-30 (Estimated); Study Completion 2026-12-28 (Estimated)

PRIMARY OUTCOMES:
Client Satisfaction Questionnaire | baseline
  The Client Satisfaction Questionnaire (CSQ) is an 8-item scale with response options ranging from 1 - 4. Total scores range from 8 -32. Higher scores indicate higher satisfaction. Assesses the extent to which parents found the intervention helpful, relevant, feasible, and effective.
Client Satisfaction Questionnaire | 11 weeks
  The Client Satisfaction Questionnaire (CSQ) is an 8-item scale with response options ranging from 1 - 4. Total scores range from 8 -32. Higher scores indicate higher satisfaction. Assesses the extent to which parents found the intervention helpful, relevant, feasible, and effective.
Parent-Patient Activation Measure - Mental Health | baseline
  The Parent-Patient Activation Measure - Mental Health measures parent activation, defined as the knowledge, ability, and confidence to manage their child's mental health care. It consists of 13 items on a 4-point Likert-type scale ranging from 1-4. Item scores are summed for a total composite score ranging from 13 -52. Composite scores are linearly transformed into scores ranging from 0 - 100. Higher scores indicate higher activation in managing their child's mental health care.
Parent-Patient Activation Measure - Mental Health | 11 weeks
  The Parent-Patient Activation Measure - Mental Health measures parent activation, defined as the knowledge, ability, and confidence to manage their child's mental health care. It consists of 13 items on a 4-point Likert-type scale ranging from 1-4. Item scores are summed for a total composite score ranging from 13 -52. Composite scores are linearly transformed into scores ranging from 0 - 100. Higher scores indicate higher activation in managing their child's mental health care.
Family Empowerment Scale | baseline
  The Family Empowerment Scale consists of 34-items and 3 subscales (1. Family, 2. Mental health services, 3. Community) designed to assess a parent's sense of empowerment in families of children with an emotional disorder. Response options range from 1 (not true at all) - 5 (very true). Total scores range from 34 - 170, with higher scores indicating higher levels of empowerment.
Family Empowerment Scale | 11 weeks
  The Family Empowerment Scale consists of 34-items and 3 subscales (1. Family, 2. Mental health services, 3. Community) designed to assess a parent's sense of empowerment in families of children with an emotional disorder. Response options range from 1 (not true at all) - 5 (very true). Total scores range from 34 - 170, with higher scores indicating higher levels of empowerment.

SECONDARY OUTCOMES:
PROMIS Parent-Proxy Pediatric Anxiety Short Form 8a (PROMIS Anxiety) | baseline
  The PROMIS Parent-Proxy Pediatric Anxiety Short Form 8a is an 8-item measure that assesses symptoms of fear, anxious misery, hyperarousal, and somatic symptoms related to arousal among pediatric populations aged 5- to 17-years old. It is a parent report with response options that range from 1 (never) to 5 (almost always). Total scores range from 8 -40 with higher scores indicating higher levels of anxiety.
PROMIS Parent-Proxy Pediatric Anxiety Short Form 8a (PROMIS Anxiety) | 11 weeks
  The PROMIS Parent-Proxy Pediatric Anxiety Short Form 8a is an 8-item measure that assesses symptoms of fear, anxious misery, hyperarousal, and somatic symptoms related to arousal among pediatric populations aged 5- to 17-years old. It is a parent report with response options that range from 1 (never) to 5 (almost always). Total scores range from 8 -40 with higher scores indicating higher levels of anxiety.
PROMIS Parent-Proxy Pediatric Depressive Symptoms Short Form 8a (PROMIS Depressive) | baseline
  The PROMIS Parent-Proxy Pediatric Depressive Symptoms Short Form 8a is an 8-item measures that assesses negative mood and views of self, social cognition, and decreased positive affect and engagement among pediatric populations aged 5- to 17-years old. It is a parent-report and response options range from 1 (never) to 5 (almost always). Total scores range from 8 - 40 with higher scores indicating higher levels of depressive symptomatology.
PROMIS Parent-Proxy Pediatric Depressive Symptoms Short Form 8a (PROMIS Depressive) | 11 weeks
  The PROMIS Parent-Proxy Pediatric Depressive Symptoms Short Form 8a is an 8-item measures that assesses negative mood and views of self, social cognition, and decreased positive affect and engagement among pediatric populations aged 5- to 17-years old. It is a parent-report and response options range from 1 (never) to 5 (almost always). Total scores range from 8 - 40 with higher scores indicating higher levels of depressive symptomatology.
Pediatric Symptom Checklist - 17 (PSC-17) | baseline
  The Pediatric Symptom Checklist - 17 (PSC-17) is a 17-item measures that assesses child psychosocial function associated with internalizing, externalizing, and attention problems in children aged 5- to 17-years old. The parent report version will be used. Response options range from 0 (Never) - 2 (Often). Total scores range from 0 - 51; Scores on the Internalizing subscale range from 0 - 15, Scores on the Attention subscale range from 0 - 15, Scores on the Externalizing subscale range from 0 - 35. Higher scores indicate higher levels of symptomatology.
Pediatric Symptom Checklist - 17 (PSC-17) | 11 weeks
  The Pediatric Symptom Checklist - 17 (PSC-17) is a 17-item measures that assesses child psychosocial function associated with internalizing, externalizing, and attention problems in children aged 5- to 17-years old. The parent report version will be used. Response options range from 0 (Never) - 2 (Often). Total scores range from 0 - 51; Scores on the Internalizing subscale range from 0 - 15, Scores on the Attention subscale range from 0 - 15, Scores on the Externalizing subscale range from 0 - 35. Higher scores indicate higher levels of symptomatology.
Barriers to Treatment Participation Scale; subscales I - IV | baseline
  The Barriers to Treatment Participation Scale consists of 44 items and 4 subscales. The subscales include: I. Stressors (20 items; Response options 1 (never a problem) -5 (very often a problem)); II. Tx Demands (10 items; Response options 1-5); III Relevance (8 items; Response options: 1-5); IV Relationship (6 items; 1 -5); Total scores for the subscales with continuous response options range from 44- 220, With higher scores indicating higher barriers to treatment participation.
Barriers to Treatment Participation Scale; subscale V | baseline
  The Barriers to Treatment Participation Scale consists of a fifth subscale, Critical Events (14 items; scored yes/no).
  Measures the extent to which the parent experienced barriers to their child participating in treatment, and specific types of barriers to treatment.
Barriers to Treatment Participation Scale; subscales I - IV | 11 weeks
  The Barriers to Treatment Participation Scale consists of 44 items and 4 subscales. The subscales include: I. Stressors (20 items; Response options 1 (never a problem) -5 (very often a problem)); II. Tx Demands (10 items; Response options 1-5); III Relevance (8 items; Response Options: 1-5); IV Relationship (6 items; 1 -5); Total scores for the subscales with continuous response options range from 44- 220, With higher scores indicating higher barriers to treatment participation.
Barriers to Treatment Participation Scale; subscale V | 11 weeks
  The Barriers to Treatment Participation Scale consists of a fifth subscale, Critical Events (14 items; scored yes/no).
  Measures the extent to which the parent experienced barriers to their child participating in treatment, and specific types of barriers to treatment.
Difficulties in Emotion Regulation Scale (DERS) | baseline
  Measures four aspects of parental emotion regulation: (a) awareness and understanding of emotions; (b) acceptance of emotions; (c) the ability to control impulses and behave in accordance with goals in the presence of negative affect; and (d) access to emotion.
Difficulties in Emotion Regulation Scale (DERS) | 11 weeks
  Measures four aspects of parental emotion regulation: (a) awareness and understanding of emotions; (b) acceptance of emotions; (c) the ability to control impulses and behave in accordance with goals in the presence of negative affect; and (d) access to emotion.

OTHER OUTCOMES:
Post-Session Items | 1 week
  There are 9 post-session items for participants and 2 post-session items for parent coaches. The post session items for participants include a mixture of likert-type items and open-ended responses to assess aspects of Acceptability, Usefulness, and Feasibility of each session. There are no total scores given. The investigators will use the information to refine the curriculum. The parent coach items assess parent coach perceptions of ability to adhere to the session plan and asking if they have any suggestions to improve the session.
Post-Session Items | 2 weeks
  There are 9 post-session items for participants and 2 post-session items for parent coaches. The post session items for participants include a mixture of likert-type items and open-ended responses to assess aspects of Acceptability, Usefulness, and Feasibility of each session. There are no total scores given. The investigators will use the information to refine the curriculum. The parent coach items assess parent coach perceptions of ability to adhere to the session plan and asking if they have any suggestions to improve the session.
Post-Session Items | 3 weeks
  There are 9 post-session items for participants and 2 post-session items for parent coaches. The post session items for participants include a mixture of likert-type items and open-ended responses to assess aspects of Acceptability, Usefulness, and Feasibility of each session. There are no total scores given. The investigators will use the information to refine the curriculum. The parent coach items assess parent coach perceptions of ability to adhere to the session plan and asking if they have any suggestions to improve the session.
Post-Session Items | 4 weeks
  There are 9 post-session items for participants and 2 post-session items for parent coaches. The post session items for participants include a mixture of likert-type items and open-ended responses to assess aspects of Acceptability, Usefulness, and Feasibility of each session. There are no total scores given. The investigators will use the information to refine the curriculum. The parent coach items assess parent coach perceptions of ability to adhere to the session plan and asking if they have any suggestions to improve the session.
Post-Session Items | 5 weeks
  There are 9 post-session items for participants and 2 post-session items for parent coaches. The post session items for participants include a mixture of likert-type items and open-ended responses to assess aspects of Acceptability, Usefulness, and Feasibility of each session. There are no total scores given. The investigators will use the information to refine the curriculum. The parent coach items assess parent coach perceptions of ability to adhere to the session plan and asking if they have any suggestions to improve the session.
Post-Session Items | 6 weeks
  There are 9 post-session items for participants and 2 post-session items for parent coaches. The post session items for participants include a mixture of likert-type items and open-ended responses to assess aspects of Acceptability, Usefulness, and Feasibility of each session. There are no total scores given. The investigators will use the information to refine the curriculum. The parent coach items assess parent coach perceptions of ability to adhere to the session plan and asking if they have any suggestions to improve the session.
Post-Session Items | 7 weeks
  There are 9 post-session items for participants and 2 post-session items for parent coaches. The post session items for participants include a mixture of likert-type items and open-ended responses to assess aspects of Acceptability, Usefulness, and Feasibility of each session. There are no total scores given. The investigators will use the information to refine the curriculum. The parent coach items assess parent coach perceptions of ability to adhere to the session plan and asking if they have any suggestions to improve the session.
Post-Session Items | 8 weeks
  There are 9 post-session items for participants and 2 post-session items for parent coaches. The post session items for participants include a mixture of likert-type items and open-ended responses to assess aspects of Acceptability, Usefulness, and Feasibility of each session. There are no total scores given. The investigators will use the information to refine the curriculum. The parent coach items assess parent coach perceptions of ability to adhere to the session plan and asking if they have any suggestions to improve the session.
Post-Session Items | 9 weeks
  There are 9 post-session items for participants and 2 post-session items for parent coaches. The post session items for participants include a mixture of likert-type items and open-ended responses to assess aspects of Acceptability, Usefulness, and Feasibility of each session. There are no total scores given. The investigators will use the information to refine the curriculum. The parent coach items assess parent coach perceptions of ability to adhere to the session plan and asking if they have any suggestions to improve the session.
Post-Session Items | 10 weeks
  There are 9 post-session items for participants and 2 post-session items for parent coaches. The post session items for participants include a mixture of likert-type items and open-ended responses to assess aspects of Acceptability, Usefulness, and Feasibility of each session. There are no total scores given. The investigators will use the information to refine the curriculum. The parent coach items assess parent coach perceptions of ability to adhere to the session plan and asking if they have any suggestions to improve the session.

CONTACTS AND LOCATIONS:
Overall Officials: Heather J Risser, PhD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
We are concerned that parents will be less likely to participate if their individual participant data is to be shared. Particularly in communities of color, there is a history of exploitation in research.

DOCUMENTS (3):
  • Study Protocol (2021-12-08): https://cdn.clinicaltrials.gov/large-docs/00/NCT04986800/Prot_003.pdf
  • Statistical Analysis Plan (2021-06-16): https://cdn.clinicaltrials.gov/large-docs/00/NCT04986800/SAP_001.pdf
  • Informed Consent Form (2020-12-15): https://cdn.clinicaltrials.gov/large-docs/00/NCT04986800/ICF_004.pdf